CLINICAL TRIAL: NCT04313140
Title: Virtual Biopsy Development to Identify Patient's Glioma Grade at the CHU of Poitiers Using Magnetic Resonance Imaging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-A02531-56
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Development of the Virtual Biopsy; Tumor Grade; Artificial Intelligence Algorithms; Clinical; Radiological
MeSH Terms: interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient's Glioma grade (Experimental): magnetic resonance spectroscopy
  Interventions: Diagnostic Test: Diagnostic test

INTERVENTIONS:
Diagnostic Test: Diagnostic test — The intervention occurs only one time (for 2h30), the MRI examination is divided as follow:
  * Cinicial MRI (50 minutes)
  * Research MRI (Phosphorus Spectroscopy, Sodium Imaging)

SUMMARY:
Glioma is a tumor of the central nervous system. These lesions are sorted with the WHO ranking regarding the tumoral oncotype. The tumoral MRI assessment is the first step before any medical decision. Currently, only anatomical biopsy can give the tumor grade definition and help to define the most adapted treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age≥ 18 years,
* Patient with suspected glioma with prior imaging
* Subject free, with legal protection guardianship or curatorship;
* Enrollment in the French Social Security system;
* Informed consent signed by the patient

Exclusion Criteria:

* Any contraindication to an MRI examination
* Legal protection, namely minors, persons deprived of their liberty by a judicial or administrative decision, persons residing in a health or social establishment, adults under legal protection and finally patients in emergency situations
* Pregnant or lactating women, women of childbearing age who do not have effective contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-02-22 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Validation of the virtual biopsy in the context of gliomas through the use of statistical learning algorithms (artificial intelligence) compared to the biopsy. | The MRI examination (for 2 hours 30 minutes)
  Evaluate the diagnostic capabilities of artificial intelligence algorithms for virtual biopsy based on sensitivity and specificity

CONTACTS AND LOCATIONS:
Locations (1):
- CHU De Poitiers, Poitiers, France